CLINICAL TRIAL: NCT04495933
Title: A Phase 1, Randomised, Double-Blind, Placebo-Controlled, Dosage-Escalation, Single Centre Study to Evaluate the Safety and Immunogenicity of an Adjuvanted SARS-CoV-2 Sclamp Protein Subunit Vaccine in Healthy Adults Aged 18 to 55 Years Old and Healthy Older Adults, Aged 56 Years and Over
Brief Title: A Study on the Safety, Tolerability and Immune Response of SARS-CoV-2 Sclamp (COVID-19) Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: Syneos Health (Other); Coalition for Epidemic Preparedness Innovations (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: UQ-1-SARS-CoV-2-Sclamp; ACTRN12620000674932p (Registry Identifier: ANZCTR)
Record Dates: First submitted 2020-07-13; First posted 2020-08-03 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2021-08

CONDITIONS: SARS-CoV2; Covid19
Keywords: SARS-CoV-2 infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Cohort 1: SARS-CoV-2 Sclamp vaccine 5 mcg, or placebo Cohort 2: SARS-CoV-2 Sclamp vaccine 15 mcg, or placebo Cohort 3: SARS-CoV-2 Sclamp vaccine 45 mcg, or placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MF59 adjuvanted SARS-CoV-2 Sclamp vaccine 5mcg (Experimental): SARS-CoV-2 Sclamp antigen 5 mcg mixed with MF59 adjuvant in 0.5 mL suspension, administered in a two dose regimen, at least 28 days apart.(Cohorts 1 & 4)
  Interventions: Biological: MF59 adjuvanted SARS-CoV-2 Sclamp vaccine 5mcg; Other: Placebo
- MF59 adjuvanted SARS-CoV-2 Sclamp vaccine 15mcg (Experimental): SARS-CoV-2 Sclamp antigen 15 mcg mixed with MF59 adjuvant in 0.5 mL suspension, administered in a two dose regimen, at least 28 days apart. (Cohorts 2 & 5)
  Interventions: Biological: MF59 adjuvanted SARS-CoV-2 Sclamp vaccine 15mcg; Other: Placebo
- MF59 adjuvanted SARS-CoV-2 Sclamp vaccine 45mcg (Experimental): SARS-CoV-2 Sclamp antigen 45 mcg mixed with MF59 adjuvant in 0.5 mL suspension, administered in a two dose regimen, at least 28 days apart. (Cohorts 3 & 6)
  Interventions: Biological: MF59 adjuvanted SARS-CoV-2 Sclamp vaccine 45mcg; Other: Placebo

INTERVENTIONS:
Biological: MF59 adjuvanted SARS-CoV-2 Sclamp vaccine 5mcg — MF59 adjuvanted SARS-CoV-2 Sclamp vaccine 5mcg
  Arms: MF59 adjuvanted SARS-CoV-2 Sclamp vaccine 5mcg
Biological: MF59 adjuvanted SARS-CoV-2 Sclamp vaccine 15mcg — MF59 adjuvanted SARS-CoV-2 Sclamp vaccine 15mcg
  Arms: MF59 adjuvanted SARS-CoV-2 Sclamp vaccine 15mcg
Biological: MF59 adjuvanted SARS-CoV-2 Sclamp vaccine 45mcg — MF59 adjuvanted SARS-CoV-2 Sclamp vaccine 45mcg
  Arms: MF59 adjuvanted SARS-CoV-2 Sclamp vaccine 45mcg
Other: Placebo — sterile saline

SUMMARY:
This study is being conducted to look at the safety and immune response (how the immune system of the human body reacts) to a vaccine for SARS-CoV-2 (the virus responsible for COVID-19 infection) when administered as an intramuscular injection (an injection directly into the muscle) to the upper arm of healthy participants, on two occasions at least 28 days apart.

DETAILED DESCRIPTION:
This study will be conducted in 2 parts: Part 1 will include a young healthy adult population aged ≥ 18 - ≤ 55 years and Part 2 will include an older healthy adult population aged 56 years and over.

The study will consist of 6 cohorts: 2 cohorts of a lower dose (Treatment A), 2 cohorts of an intermediate dose (Treatment B) and 1 cohort of a higher dose (Treatment C) (Part 2 only), and 1 cohort of a higher dose examining both a two dose regimen (Treatment C) and a single dose vaccination regimen (Treatment D) (Part 1 only).

Cohorts 1,2 and 3 will include subjects aged ≥ 18 - ≤ 55 years of age and cohorts 4, 5 and 6 will include subjects aged 56 years and older. Cohorts 4, 5 and 6 will include an approximately equal number of subjects aged ≥ 56 - ≤ 65 years of age, and ≥ 66 years and over.

Part 1: Cohort 1 will include 32 subjects; of these 8 will receive placebo, and 24 subjects will receive Treatment A. Cohort 2 will include 32 subjects; of these 8 will receive placebo, and 24 subjects will receive Treatment B. Cohort 3 will include 56 subjects; of these 8 will receive placebo, 24 subjects will receive Treatment C, and 24 subjects will receive Treatment D.

Part 2: Cohort 4 will include 32 subjects; of these 8 will receive placebo, and 24 subjects will receive Treatment A. Cohort 5 will include 32 subjects; of these 8 will receive placebo, and 24 subjects will receive Treatment B. Cohort 6 will include 32 subjects; of these 8 will receive placebo, and 24 subjects will receive Treatment C.

Sentinels will be used for each cohort in Part 1 such that the first two subjects will receive either the first dose of SARS-CoV-2 Sclamp vaccine or placebo. After at least 24 hours from the time of administration of the first doses a review of the immediate post-vaccination safety data will be conducted by the Safety Review Committee (SRC) in accordance with the study protocol. Should there be no safety concerns, the remaining participants in each cohort will be dosed. The step-wise dose escalation study design is an additional precautionary measure, where the lower dose cohort will complete their first vaccination, and the cumulative safety data from the first 7 days will be evaluated by the SRC prior to initiating vaccination with the next higher dose of vaccine.

Cohorts will be dosed sequentially, and escalation from Cohort 1 to Cohort 3 will be authorised by the SRC if no safety events of concern are observed in subjects up to Day 8 following review of the cumulative safety data of each Cohort.

After the first vaccination dose has been administered to Cohorts 1, 2 and 3 and the aggregated safety data reviewed by the SRC, vaccination will be initiated for Cohorts 4, 5 and 6. These Cohorts will not include sentinels, however, the SRC will review the aggregated/cumulative safety and tolerability data up to at least Day 8 post vaccination for all subjects in each of Cohorts 4, 5 and 6 by cohort before proceeding to the second vaccination dose.

Subjects will receive two single intramuscular (IM) doses of the following study treatments at 28 days apart as follows:

IM administration (to the deltoid region of the subjects non dominant arm, administered by a registered nurse [RN]) of SARS-CoV-2 Sclamp adjuvanted vaccine, administered on Days 1 and 29, of one of the following treatments:

Treatment A (Cohorts 1 & 4): SARS-CoV-2 Sclamp vaccine 1 x 5 mcg in 0.5 mL suspension, administered as two separate doses at least 28 days apart Treatment B (Cohorts 2 & 5): SARS-CoV-2 Sclamp vaccine 1 x 15 mcg in 0.5 mL suspension, administered as two separate doses , at least 28 days apart Treatment C (Cohorts 3 & 6): SARS-CoV-2 Sclamp vaccine 1 x 45 mcg in 0.5 mL suspension, administered as two separate doses at least 28 days apart Treatment D (Cohort 3 only): SARS-CoV-2 Sclamp vaccine 1 x 45 mcg in 0.5 mL suspension, followed by placebo administered as the second dose at least 28 days apart.

The proposed escalation scheme for the study consists of two three-fold dose increments. The planned dose range of 5 mcg to 15 mcg to 45 mcg administered 28 days apart was selected to minimize the risk to the subjects while ensuring the evaluation of an exposure range that encompasses and exceeds the expected level to achieve an immunological response.

The SRC will be responsible for the assessment of available safety and tolerability data for each cohort and to make decisions with regards to study progression.

The study will be unblinded prior to Day 394. All subjects that received an investigational vaccine product (not placebo) will be offered to return for optional annual follow-up visits beyond Day 394 to determine the duration of the HIV diagnostic cross-reactivity. Samples from this visit will be tested for cross-reaction in HIV point of care and rapid diagnostic tests.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female, ≥18 and ≤55 years of age, with BMI >18 and <34.0 kg/m2 and body weight ≥50.0 kg for males and ≥45.0 kg for females (Part 1); Healthy male or non-pregnant female, ≥56 years of age, with BMI >18 and <34.0 kg/m2 and body weight ≥50.0 kg for males and ≥45.0 kg for females (Part 2)
* Healthy as defined by:

  1. The absence of clinically significant illness and surgery within 28 days prior to dosing. Subjects displaying signs or symptoms of an acute and/or febrile illness within 24 hours pre-dose (with at least 3 symptom-free pre-dose days required) will be carefully evaluated for upcoming illness/disease. Inclusion pre-dosing is at the discretion of the Investigator, and the subject may have their scheduled dosing postponed until the condition resolves.
  2. The absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, haematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease (Part 1); b. The absence of clinically significant history of a pre-existing medical condition that is not stable (neurological, endocrine, cardiovascular, respiratory, haematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease). A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months before enrolment (Part 2)
* Non-smokers or social smokers (defined as the equivalent of fewer than 10 cigarettes per week). Ex-heavy smokers (heavy smoking defined as the equivalent of 25 or more cigarettes per day) may be admitted if they have quit, or reduced their cigarette intake to the defined level of social smoking, for a period of at least 12 months.
* Women of childbearing potential (WOCBP) or men whose sexual partners are WOCBP must be able and willing to use at least 2 highly effective methods of contraception commencing at enrolment, during the study and for 3 months after last treatment administration. A female subject is considered to be a WOCBP following menarche and until she is in a postmenopausal state for 12 consecutive months (without an alternative medical cause) or otherwise permanently sterile (for which acceptable methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy). A follicle-stimulating hormone (FSH) test may be used to confirm post-menopausal state. Examples of acceptable methods of contraceptive methods (for female subjects) to be used throughout the study include:

  1. Simultaneous use of hormonal contraceptives, started at least 28 days prior to first study treatment administration and must agree to use the same hormonal contraceptive throughout the study, and condom for the male partner;
  2. Simultaneous use of intra-uterine contraceptive device, placed at least 28 days prior to first study treatment administration, and condom for the male partner;
  3. Simultaneous use of diaphragm or cervical cap and male condom for the male partner, started at least 28 days prior to first study treatment administration;
  4. Sterile male partner (vasectomized since at least 6 months prior to first study treatment administration);
  5. True abstinence, defined as no sexual intercourse with a male partner, (for heterosexual couples) for at least 28 days prior to first study treatment administration and for at least the duration of the study. Periodic abstinence and withdrawal are not acceptable methods.
* WOCBP must have a negative urine pregnancy test prior to receiving each dose.
* Male subjects (including men who have had a vasectomy) with a pregnant partner, a female partner not of childbearing potential, or a same sex partner, must agree to use a condom from the first study treatment administration until at least 90 days after the last study treatment administration.
* Male subjects must be willing not to donate sperm until 90 days following the last study treatment administration.
* Must be able to attend all visits for the duration of the study and to comply with all study procedures according to the study schedule.
* Capable of, and have given, written informed consent.

Exclusion Criteria:

* Any clinically significant abnormality or vital sign abnormality at physical examination (including baseline high blood pressure [140/90] after 3 repeated measurements or high random blood sugar [non-fasting]), clinically significant abnormal laboratory test results or positive test for HIV, hepatitis B, or hepatitis C found during medical screening (Part 1); Any clinically significant abnormality or vital sign abnormality at physical examination, or uncontrolled hypertension in adults aged ≥ 56 years and older ,or high random blood sugar [non-fasting]), clinically significant abnormal laboratory test results or positive test for HIV, hepatitis B, or hepatitis C found during medical screening (Part 2).
* Any acute or chronic ongoing illness which, in the judgement of the investigator, may preclude the subject's participation.
* Any subject that has an active COVID-19 infection (positive COVID-19 test: nasal/oropharyngeal swab and/or positive serum antibody response) at screening, or Day 1, or has been in close contact with someone who has an active COVID-19 infection, or has recovered from a previous COVID-19, SARS-CoV-1, or MERS infection.
* Positive pregnancy, urine drug screen, or alcohol breath test at screening.
* Known history of allergic reactions or hypersensitivity to vaccines, or to any excipient in the formulation (including the adjuvant, MF59C.1).
* Presence of a known, or suspected, impairment of the immune system including, but not limited to, HIV, autoimmune disorders, immunosuppressant therapy, and diabetes mellitus.
* History of a known, or suspected, respiratory system disorder including, but not limited to, cystic fibrosis, reactive airway disease, emphysema, chronic bronchitis, chronic obstructive pulmonary disease (COPD), or asthma, excluding childhood asthma (Part 1); History of a known, or suspected, or currently unstable medical condition that may expose the participant to an increased risk for severe SARS-CoV-2 disease, such as a respiratory system disorder including, but not limited to, cystic fibrosis, reactive airway disease, emphysema, chronic bronchitis, chronic obstructive pulmonary disease (COPD), or asthma, excluding childhood asthma, uncontrolled hypertension, ischemic or structural heart disease, chronic kidney disease, chronic liver disease, endocrine disorder and neurological illness (Part 2).
* History of significant alcohol abuse within 12 months prior to screening.
* Positive test for drugs of abuse (such as marijuana/tetrahydrocannabinol [THC] products, amphetamine, methamphetamine, methadone, barbiturates, benzodiazepines, cocaine, opiates, methylenedioxymethamphetamine [MDMA], or phencyclidine [PCP]) at screening, prior to dosing, or a history of drug abuse within 12 months prior to screening.
* Participation in a clinical research study involving the administration of an investigational, or marketed, drug or device within 30 days prior to receiving the first treatment administration, or administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug, vaccine, or device administration, or intent to participate in another clinical study at any time during the conduct of the study.
* Use of medications for the timeframes specified below, with the exception of hormonal contraceptives and medications exempted by the Investigator on a case-by-case basis because they are judged to interfere with subject safety e.g., topical drug products without significant systemic absorption are permissible:

  1. Prescription medication within 14 days prior to the first dosing (Part 1); Prescription medication within 14 days prior to the first dosing that in the opinion of the Investigator could impact the subjects safe participation in the study (Part 2)
  2. Any medication, or treatments, that may affect the immune system such as allergy injections, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or other drugs known to be frequently associated with significant major organ toxicity within 90 days prior to enrolment;
  3. Any registered vaccine administered within 30 days prior to enrolment in the study, or who plan to receive any non-study vaccines within 28 days of the second dose of the study vaccine
  4. Any other investigational coronavirus vaccine i.e. SARS-CoV-1, SARS-CoV-2, MERS etc. at any time prior to, or during, the study.
  5. Over-the-counter products within 7 days prior to the first dosing, with the exception of the occasional use of paracetamol (up to 2 g daily) and standard dose vitamins (Part 1); Over-the-counter products within 7 days prior to the first dosing, that in the opinion of the investigator could impact the subjects safe participation in the study. Paracetamol (up to 2 g daily) and standard dose vitamins will be permitted (Part 2).
* Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing.
* Receipt of blood products within 2 months prior to the first study treatment administration (Day 1), or planned receipt of blood products during the study period.
* Breast-feeding subject, or subject who plans to breastfeed from the time of first dose through 60 days after last study treatment administration.
* Presence of tattoos, scarring, skin discoloration, or any other skin disturbances at the injection site which, in the opinion of the Investigator, may inhibit the ability to effectively perform an injection site assessment.
* Employee or immediate relative of an employee of the clinical site, any of its affiliates or partners, or Syneos Health.
* Any reason which, in the opinion of the Investigator, would interfere with the primary study objectives or prevent the subject from participating in the study.
* Permanent resident in an aged care facility (nursing or aged care home) (Part 2 only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Frequency of Solicited local reactogenicity adverse events (AEs) | 7 days following each vaccination (at Days 1 and 29)
  - the frequency of solicited local reactogenicity adverse events (AEs)
Frequency of Solicited systemic reactogenicity adverse events (AEs) | 7 days following each vaccination (at Days 1 and 29)
  - the frequency of solicited systemic reactogenicity AEs
Grading of Solicited local reactogenicity adverse events (AEs) | 7 days following each vaccination (at Days 1 and 29)
  - the grading of solicited local reactogenicity adverse events (AEs)
Grading of Solicited systemic reactogenicity adverse events (AEs) | 7 days following each vaccination (at Days 1 and 29)
  - the grading of solicited systemic reactogenicity AEs
Unsolicited adverse events (AEs) | 28 days following each vaccination (at Days 1 and 29)
  - the frequency, duration, intensity and relationship to vaccination of unsolicited local adverse events (AEs)
Serious adverse events (SAEs), Medically attended adverse events (MAAEs) and any Adverse events (AEs) leading to study withdrawal at any time during the study | through study completion (394 days)
  - the frequency, duration, intensity and relationship to vaccination of Serious adverse events (SAEs), Medically attended adverse events (MAAEs) and any Adverse events (AEs) leading to study withdrawal at any time during the study (including decision by the Principal Investigator [PI] not to proceed with the second dose) at any time during the study
Geometric Mean Titer (GMT) of the serum antibody response | 28 days following each vaccination (Days 29 and 57)
  - Geometric mean titre (GMT) of the serum antibody response compared to placebo
Geometric Mean Titer (GMT) of the serum neutralizing antibody (NAb) response to SARS-CoV-2 virus | 28 days following each vaccination (Days 29 and 57)
  GMT of the serum NAb titres to SARS-CoV-2 virus compared to placebo

SECONDARY OUTCOMES:
Total serum antibody immune responses | through study completion (394 days)
  GMT of the serum antibody response compared to placebo
proportion of participants with ≥ 4 fold increase in titer above baseline | through study completion (394 days)
  proportion of participants with greater than or equal to 4 fold increase in titre above baseline compared to placebo.
GMT of the serum neutralizing antibody (NAb) titres | through study completion (394 days)
  GMT of the serum neutralizing antibody (NAb) immune responses compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Paul Griffin, Dr, Principal Investigator — Nucleus Network Brisbane
Locations (1):
- Nucleus Network Brisbane (Q-Pharm Pty Ltd), Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Yes
individual participant data underlying published results only on a case-by-case basis at the discretion of Primary Sponsor
Supporting Information: CSR
Time Frame: Immediately following publication, no end date
Access Criteria: Available only to achieve the aims in the approved proposal

REFERENCES:
- [Derived] Chappell KJ, Mordant FL, Amarilla AA, Modhiran N, Liang B, Li Z, Wijesundara DK, Lackenby JA, Griffin P, Bennet JK, Hensen L, Zhang W, Nguyen THO, Tran MH, Tapley P, Barnes J, Reading PC, Kedzierska K, Ranasinghe C, Subbarao K, Watterson D, Young PR, Munro TP. Long-term safety and immunogenicity of an MF59-adjuvanted spike glycoprotein-clamp vaccine for SARS-CoV-2 in adults aged 18-55 years or >/=56 years: 12-month results from a randomised, double-blind, placebo-controlled, phase 1 trial. EBioMedicine. 2023 Nov;97:104842. doi: 10.1016/j.ebiom.2023.104842. Epub 2023 Oct 20. PMID 37865043
- [Derived] Chappell KJ, Mordant FL, Li Z, Wijesundara DK, Ellenberg P, Lackenby JA, Cheung STM, Modhiran N, Avumegah MS, Henderson CL, Hoger K, Griffin P, Bennet J, Hensen L, Zhang W, Nguyen THO, Marrero-Hernandez S, Selva KJ, Chung AW, Tran MH, Tapley P, Barnes J, Reading PC, Nicholson S, Corby S, Holgate T, Wines BD, Hogarth PM, Kedzierska K, Purcell DFJ, Ranasinghe C, Subbarao K, Watterson D, Young PR, Munro TP. Safety and immunogenicity of an MF59-adjuvanted spike glycoprotein-clamp vaccine for SARS-CoV-2: a randomised, double-blind, placebo-controlled, phase 1 trial. Lancet Infect Dis. 2021 Oct;21(10):1383-1394. doi: 10.1016/S1473-3099(21)00200-0. Epub 2021 Apr 19. PMID 33887208

DOCUMENTS (1):
  • Study Protocol (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT04495933/Prot_000.pdf